CLINICAL TRIAL: NCT05783843
Title: Comparison of Text and Pictorial Waterpipe Tobacco Warnings Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00091946; R01CA241420 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-24 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-03

CONDITIONS: Waterpipe Tobacco Smoking
Keywords: Waterpipe Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Participants randomized to the text-only condition will see six packages with different text warnings. Participants randomized to the pictorial condition will see six packages with different pictorial warnings. Participants in the control condition will see a single package without a warning.
Who Masked: Participant
Masking Description: Participants will be blinded as to the comparators for their arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pictorial Warnings (Experimental): Waterpipe tobacco packages shown with pictorial warnings about health harms of waterpipe smoking
  Interventions: Behavioral: Pictorial Warnings
- Text Warnings (Experimental): Waterpipe tobacco packages shown with text-only warning about health harms of waterpipe smoking
  Interventions: Behavioral: Text Warnings
- No Warnings (Control) (Experimental): Waterpipe tobacco package shown without a warning
  Interventions: Behavioral: No Warnings (Control)

INTERVENTIONS:
Behavioral: Pictorial Warnings — Participants will be shown 6 waterpipe tobacco packages with 6 different pictorial warnings about the health harms of waterpipe smoking. The order of the 6 packages within this trial arm will be randomized. Study investigators developed a fictitious waterpipe tobacco brand to be used in this study and designed the warnings for this arm.
  Arms: Pictorial Warnings
Behavioral: Text Warnings — Participants will be shown 6 waterpipe tobacco packages with 6 different text-only warnings about the health harms of waterpipe smoking. The order of the 6 packages within this trial arm will be randomized. Study investigators developed a fictitious waterpipe tobacco brand to be used in this study and designed the warnings for this arm.
  Arms: Text Warnings
Behavioral: No Warnings (Control) — Participants will be shown a single package without a warning. Study investigators developed a fictitious waterpipe tobacco brand to be used in this study.
  Arms: No Warnings (Control)

SUMMARY:
The purpose of this study is to whether exposure to waterpipe tobacco warnings reduce young adults' intentions to smoke waterpipe in the future.

DETAILED DESCRIPTION:
Young adults, defined as those 18-29 years old, have the highest rates of waterpipe tobacco smoking, which increases their risk of a variety of pulmonary, neurological, and oncological health conditions, among many others. This trial will randomly assign young adult waterpipe users or those susceptible to use to view waterpipe tobacco packages with text warning, pictorial warnings, or no warnings in a one-time online study. Participants will answer a series of questions regarding each package.

ELIGIBILITY:
Inclusion Criteria:

* United States (US) Resident
* Has used waterpipe tobacco within the past year (self-report) OR
* Has not used waterpipe tobacco within the past year but is susceptible to use (self-report)

Exclusion Criteria:

* Younger than 18 or older than 29
* Not a US Resident
* Has not used waterpipe tobacco within the past year and is not susceptible to use (self-report)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1215 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Sutfin, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Warnings | Pictorial Warnings | No Warnings (Control)
Started | 396 | 402 | 417
Completed | 396 | 402 | 417
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Warnings | Pictorial Warnings | No Warnings (Control) | Total
Number analyzed (Participants) | 396 | 402 | 417 | 1215
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3.2) | 24.9 (3.4) | 25 (3.3) | 25 (3.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 253 | 270 | 266 | 789
  Male | 143 | 131 | 151 | 425
  Unknown/Not Reported | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 86 | 77 | 264
  Not Hispanic or Latino | 295 | 316 | 340 | 951
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 6 | 11
  Asian | 25 | 33 | 26 | 84
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 82 | 92 | 97 | 271
  White | 219 | 236 | 234 | 689
  More than one race | 34 | 18 | 30 | 82
  Unknown or Not Reported | 32 | 21 | 23 | 76
Region of Enrollment [Number; unit: participants]
  United States | 396 | 402 | 417 | 1215

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Intentions
Description: The primary outcome is intention to smoke tobacco in a waterpipe within the next year, measured by averaging three items to create a composite score (adapted from research on cigarette smoking). The primary outcome will be measured after the exposure to waterpipe packages. Score ranges from 1-5 with higher score indicating greater intention to smoke hookah.
  1. How interested are you in smoking hookah in the next year?
  2. How likely are you to smoke hookah in the next year?
  3. How much do you plan to smoke hookah in the next year? Response scale: (1) Not at all / (2) Very little / (3) Somewhat / (4) Quite a bit / (5) Very interested/likely/much
Time Frame: Minute 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Text Warnings | Pictorial Warnings | No Warnings (Control)
Number analyzed (Participants) | 396 | 402 | 417
score on a scale | 1.83 (0.07) | 1.72 (0.05) | 2.21 (0.07)

2. Other Pre Specified Outcome: Product Appeal
Description: Three items will be used to measure how appealing each waterpipe tobacco package is to respondents, how likely they would be to try the product, and how much the packaging makes the respondent think that the product is harmful.
  1. How appealing is this product to you?
  2. How likely would you be to try this product?
  3. How much does this packaging make you think this product is harmful? Response scale: (1) Not at all / (2) A little / (3) Somewhat / (4) A lot
Time Frame: Minute 2
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Perceived Message Effectiveness
Description: This outcome will be measured using the 3-item Perceived Measured Effectiveness scale created by Noar and colleagues that includes items on attitudes, risk beliefs, and intentions. Mean scores will be calculated.
  1. How much does this warning make smoking hookah seem unpleasant to you?
  2. How much does this warning make you concerned about the health effects of smoking hookah?
  3. How much does this warning discourage you from wanting to smoke hookah? Response scale: (1) Not at all / (2) Very little / (3) Somewhat / (4) Quite a bit / (5) A great deal
Time Frame: Minute 2
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Attention
Description: One item to measure self-reported attention to the warning.
  1. How much does this warning grab your attention? Response scale: (1) Not at all / (2) Very little / (3) Somewhat / (4) Quite a bit / (5) A great deal
Time Frame: Minute 1
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Emotional Reactions
Description: Three items to measure negative emotional reactions to the warning that the participant saw. Mean scores will be calculated.
  1. How much does this warning make you feel anxious?
  2. How much does this warning make you feel disgusted?
  3. How much does this warning make you feel scared? Response scale: (1) Not at all / (2) Very little / (3) Somewhat / (4) Quite a bit / (5) A great deal
Time Frame: Minute 2
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cognitive Elaboration
Description: One item to measure the extent to which a participant reports the warning making them think about the risks of hookah smoking.
  1. How much does this warning make you think about the health effects of smoking hookah? Response scale: (1) Not at all / (2) Very little / (3) Somewhat / (4) Quite a bit / (5) A great deal
Time Frame: Minute 1
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Self-reported Learning
Description: One item to measure the extent to which respondents learned something new from the warning.
  1. To what extent did you learn something new from this warning that you did not already know? Response Scale: (1) Not at all / (2) Very little / (3) Somewhat / (4) Quite a bit / (5) A great deal
Time Frame: Minute 1
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Social Interactions
Description: One item to measure self-reported likelihood of discussing the warning shown with one's social contacts within the week following the survey.
  1. How likely are you to talk about this warning with others in the next week? Response Scale: (1) Not at all / (2) Very little / (3) Somewhat / (4) Quite a bit / (5) A great deal
Time Frame: Minute 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Knowledge
Description: Six items to measure knowledge of the potential health harms described by the warnings.
  1. Hookah smoking causes heart damage.
  2. Hookah smoking causes lung damage.
  3. Hookah smoking causes mouth cancer.
  4. Hookah smoking causes carbon monoxide poisoning.
  5. Hookah smoking during pregnancy stunts fetal growth.
  6. Hookah smoking causes nicotine addiction. Response scale: (1) True / (2) False / (3) I don't know
Time Frame: Minute 3
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Beliefs
Description: Five items to measure the respondent's belief of their own risk of experiencing each of the warning health harms. One item measures risk to pregnant people, rather than the self, since this item will be administered to all participants.
  1. If I smoke hookah, I will damage my heart.
  2. If I smoke hookah, I will damage my lungs.
  3. If I smoke hookah, I will get mouth cancer.
  4. If I smoke hookah, I will get carbon monoxide poisoning.
  5. If a person smokes hookah during pregnancy, it will stunt fetal growth.
  6. If I smoke hookah, I will become addicted. Response scale: (1) Strongly disagree / (2) Somewhat disagree / (3) Neither disagree nor agree / (4) Somewhat agree / (5) Strongly agree
Time Frame: Minute 3
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Worry
Description: Five/six items measuring a respondent's concern about their risk of warning health effects. Damage to fetuses will only be asked of respondents who report female sex at birth.
  1. If you smoke hookah, how much would you worry about getting mouth cancer?
  2. If you smoke hookah, how much would you worry about damaging your heart?
  3. If you smoke hookah, how much would you worry about damaging your lungs?
  4. If you smoke hookah, how much would you worry about getting carbon monoxide poisoning?
  5. If you smoke hookah, how much would you worry about stunting fetal growth, if you were pregnant?
  6. If you smoke hookah, how much would you worry about becoming addicted? Response scale: (1) Not at all / (2) A little / (3) Somewhat / (4) A lot
Time Frame: Minute 3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Quit Motivation
Description: Participants who report past-year use will report, on a scale of 1-10, how motivated they are to quit smoking hookah.
Time Frame: Minute 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of consent up to four weeks
Description: Participants were randomized to one of three arms; two intervention arms and one control. Participants in the intervention arm saw six fictional hookah packages with either a text-only or pictorial health warnings; control participants saw single fictional hookah tobacco package with no health warnings.
Arm/Group | Text Warnings | Pictorial Warnings | No Warnings (Control)
All-Cause Mortality (participants affected / at risk) | 0/396 | 0/402 | 0/417
Serious Adverse Events (participants affected / at risk) | 0/396 | 0/402 | 0/417
Other Adverse Events (participants affected / at risk) | 0/396 | 0/402 | 0/417

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT05783843/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT05783843/ICF_000.pdf